CLINICAL TRIAL: NCT00004122
Title: A National Phase II Trial of Intron (Interferon-alfa 2b) Plus BCG for Treatment of Superficial Bladder Cancer
Brief Title: BCG Plus Interferon Alfa 2b in Treating Patients With Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067348; RPCI-DS-99-07; NCI-G99-1605
Record Dates: First submitted 1999-12-10; First posted 2004-05-21 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Bladder Cancer
Keywords: stage I bladder cancer; recurrent bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — BCG Vaccine; Interferon-alpha

INTERVENTIONS:
Biological: BCG vaccine
Biological: recombinant interferon alfa

SUMMARY:
RATIONALE: Biological therapies such as BCG use different ways to stimulate the immune system and stop cancer cells from growing. Interferon alfa may interfere with the growth of cancer cells. Combining these therapies may be an effective treatment for bladder cancer.

PURPOSE: Phase II trial to study the effectiveness of BCG plus interferon alfa 2b in treating patients who have bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of BCG combined with interferon alfa 2b in patients with superficial bladder cancer. II. Determine the relative local and systemic toxicities of this regimen and its effect on quality of life in these patients. III. Evaluate the effect of BCG dose reduction during therapy on symptom tolerance and ability to maintain an extended treatment plan in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prior BCG exposure and BCG tolerance (no prior BCG exposure vs prior BCG exposure, BCG tolerant vs prior BCG and interferon alfa treatment failure, BCG intolerant). Patients receive induction therapy consisting of varying strengths of BCG plus interferon alfa intravesically weekly for 6 weeks. Patients with disease recurrence which is resectable and/or amenable to intravesical therapy following the first induction course may receive an additional course of induction therapy. At 3 months, patients undergo evaluatory cystoscopy and cytology. At 4 months, patients with no evidence of disease receive varying strengths of maintenance therapy consisting of BCG and interferon alfa intravesically weekly for 3 weeks. Treatment repeats every 6 months for 3 courses. Quality of life is assessed within 1 week following the last induction and maintenance treatment and prior to cystoscopy. Patients are followed every 3 months for 6 months, every 6 months for 1.5 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 660 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven transitional cell carcinoma of the bladder No muscle invasive bladder cancer, transitional cell carcinoma of the upper tract, or disease within the prostatic stroma No prior evidence of metastatic transitional cell carcinoma Prior definitive resection by partial cystectomy, nephroureterectomy, or prostatectomy allowed if current disease is limited to superficial disease of the bladder only No evidence of gross hematuria within the past 2 days

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No other active malignancies or health conditions that would preclude study No serious infection within 1 month of study No evidence of active tuberculosis No significant medical or psychiatric condition that would prevent compliance Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior intravesical interferon alfa and/or BCG At least 2 years since prior immunotherapy for other malignancies or nonmalignancies Chemotherapy: At least 4 weeks since prior intravesical chemotherapy At least 2 years since prior chemotherapy for other malignancies or nonmalignancies No concurrent cytotoxic chemotherapy for other malignancies or nonmalignancies Endocrine therapy: Not specified Radiotherapy: At least 2 years since prior pelvic radiotherapy for other malignancies or nonmalignancies No concurrent pelvic radiotherapy for other malignancies or nonmalignancies Surgery: See Disease Characteristics At least 3 weeks since prior papillary or solid transitional cell carcinoma resection, bladder biopsy, or transurethral resection of the prostate At least 4 weeks since prior surgery Other: At least 2 years since any prior cytotoxic agents for other malignancies or nonmalignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07; Primary Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Corral, MD, Study Chair — Triangle Urological Group
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States